CLINICAL TRIAL: NCT07325838
Title: The Effect of a Digital Self-Management Education and Support Program on Self-Management, Glycemic Control, and Distress in Young Adults With Type 2 Diabetes Mellitus
Brief Title: Digital Self-Management Education and Support for Young Adults With Type 2 Diabetes (DSMESYAT2DM)
Acronym: DSMESYAT2DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Turan (Other Government)
Responsible Party: Sponsor-Investigator, Recep Turan, Internal Medicine Nurse, Principal Investigator, Antalya Training and Research Hospital
Organization: Antalya Training and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSMES-2025; TBAEK-1079 (Other: AKDENIZ UNIVERSITY)
Record Dates: First submitted 2025-12-18; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Diabetes-related Distress; Diabetes Distress
Keywords: Type 2 Diabetes Mellitus; Young Adults; Diabetes Self-Management; Self-Management Education; Digital Health; eHealth; mHealth; Telehealth; Nurse-Led Intervention; Diabetes Distress; Glycemic Control; HbA1c; DSMES (Diabetes Self-Management Education and Support); Diabetes Education; Randomized Controlled Trial; Behavioral Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A single-center, parallel-group, randomized controlled trial with two arms (intervention and active control). Eligible young adults with Type 2 Diabetes Mellitus will be randomized in a 1:1 ratio, stratified by baseline HbA1c level, to receive either a 12-week nurse-led digital DSMES program or usual care with access to standard digital education materials.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to their group assignment and will be informed only that they are taking part in a study comparing two types of digital support for Type 2 Diabetes Mellitus. The investigator responsible for statistical analysis and the outcomes assessor will receive de-identified data with coded group labels and will remain unaware of the actual group allocation until all primary analyses are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-Led Digital DSMES Program (Experimental): A 12-week nurse-led digital Diabetes Self-Management Education and Support (DSMES) program delivered via a digital platform. The program is structured according to the ADCES7™ self-care behaviors and includes educational modules, self-monitoring and goal-setting tools, reminders, motivational messages, and interactive communication with a diabetes nurse and, when needed, other members of the multidisciplinary team.
  Interventions: Behavioral: Digital Nurse-Led DSMES Program
- Usual Care Plus Standard Digital Education (Active Comparator): Participants will receive usual diabetes care provided in the endocrinology clinic together with access to standard digital written diabetes education materials (for example, a nationally approved Type 2 Diabetes Mellitus patient education brochure in PDF format) via the same digital platform. Participants will be able to enter and view basic self-monitoring data but will not receive the structured nurse-led DSMES intervention or interactive counseling.
  Interventions: Behavioral: Usual Care Plus Standard Digital Education

INTERVENTIONS:
Behavioral: Digital Nurse-Led DSMES Program — A 12-week nurse-led digital Diabetes Self-Management Education and Support (DSMES) intervention delivered via a web-based and/or mobile platform. The intervention includes structured educational content based on ADCES7™ self-care behaviors, digital tools for self-monitoring and goal setting, automated reminders, motivational messages, and two-way communication with a diabetes nurse, with referral to other team members (e.g., dietitian, physician) when needed.
  Other Names: Digital DSMES
  Arms: Nurse-Led Digital DSMES Program
Behavioral: Usual Care Plus Standard Digital Education — Usual diabetes care provided at the endocrinology clinic along with access to standard digital written Type 2 Diabetes Mellitus patient education materials (e.g., a nationally approved T2DM patient education brochure in PDF format) on the digital platform. Participants can enter and view basic self-monitoring data but do not receive the structured nurse-led DSMES or individualized digital counseling.
  Arms: Usual Care Plus Standard Digital Education

SUMMARY:
This randomized controlled trial will evaluate the effect of a nurse-led digital self-management education and support program on self-management behaviors, glycemic control, and diabetes-related distress in young adults with Type 2 Diabetes Mellitus (T2DM).

Young adults with T2DM often have difficulty maintaining good glycemic control and following self-management recommendations. Digital tools and remote education may help support their daily self-care, but there is limited evidence for structured, nurse-led digital programs in this age group.

In this study, 72 young adults aged 18 to 45 years with T2DM will be recruited from the Endocrinology and Metabolism outpatient clinic of Van Regional Training and Research Hospital. Participants who meet the inclusion criteria and provide informed consent will be randomly assigned to either the intervention group or the active control group (36 participants in each group). Randomization will be stratified by baseline HbA1c level.

The intervention group will receive a 12-week nurse-led Digital Diabetes Self-Management Education and Support (DSMES) program delivered via a digital platform. The program will be based on the ADCES7™ self-care behaviors and will include structured educational modules, self-monitoring and goal-setting tools, reminders, motivational messages, and interactive communication with a diabetes nurse and, when needed, other members of the multidisciplinary team.

The active control group will receive usual diabetes care and access to standard digital written education materials (for example, the Ministry of Health Type 2 Diabetes Mellitus patient education brochure in PDF format) via the same platform, as well as basic data entry tools for tracking glucose and related information. However, they will not receive the structured nurse-led DSMES intervention.

Primary outcomes will include changes in diabetes self-management behaviors and glycemic control (for example, HbA1c) from baseline to the end of the 12-week intervention. Secondary outcomes will include changes in diabetes-related distress and user satisfaction and usability of the digital program. Data will be collected using validated questionnaires and clinical laboratory results obtained from the hospital records.

The findings of this study may provide evidence on the effectiveness of a nurse-led digital DSMES program in improving self-management, glycemic control, and distress among young adults with T2DM and may support the integration of digital education and support into routine diabetes care.

DETAILED DESCRIPTION:
Young adults with Type 2 Diabetes Mellitus (T2DM) face unique challenges related to lifestyle, work, social life, and adherence to treatment recommendations. Many patients in this age group have difficulty sustaining diabetes self-management behaviors, achieving glycemic targets, and coping with diabetes-related emotional burden. Digital health technologies offer new opportunities to provide flexible, individualized, and continuous self-management education and support. However, there is still limited evidence on structured, nurse-led digital Diabetes Self-Management Education and Support (DSMES) programs specifically designed for young adults with T2DM.

This study is a single-center, parallel-group, randomized controlled trial designed to evaluate the effectiveness of a nurse-led digital DSMES program on self-management behaviors, glycemic control, and diabetes-related distress in young adults with T2DM. The study will be conducted in the Endocrinology and Metabolism outpatient clinic of Van Regional Training and Research Hospital.

A total of 72 participants aged 18 to 45 years with a diagnosis of T2DM will be included. Eligible patients will be literate, have access to the internet and a digital device (such as a smartphone, tablet, or computer), and will not have communication barriers or major physical or mental conditions that prevent participation. Patients with Type 1 diabetes, gestational diabetes, or advanced visual impairment (for example, severe diabetic retinopathy with significant vision loss) will be excluded. After obtaining informed consent, participants will be stratified by baseline HbA1c level (for example, 6.5-9% and >9%) and then randomly assigned to either the intervention group or the active control group in a 1:1 ratio (36 participants per group). The randomization will be computer-based and performed by a researcher who is not involved in outcome assessment.

The intervention group will receive a 12-week nurse-led digital DSMES program delivered through a web-based and/or mobile digital platform. The content of the program will be structured according to the ADCES7™ self-care behaviors (healthy eating, being active, taking medication, monitoring, reducing risks, healthy coping, and problem solving). The program will include:

digital educational modules presented in text, visual, and/or video formats, tools for self-monitoring of blood glucose and other relevant parameters, individualized goal-setting and progress-tracking features, reminders and motivational messages, interactive communication with a diabetes nurse via messaging or other digital communication functions, and referral or consultation with other members of the multidisciplinary team (such as a dietitian or physician) when necessary.

The nurse will follow a structured protocol for providing education, answering questions, reinforcing self-management behaviors, and supporting problem solving and coping during the 12-week intervention period.

The active control group will receive usual diabetes care provided by the clinic and access to standard digital written diabetes education materials through the same platform. This may include nationally approved patient education brochures for T2DM (for example, the Ministry of Health Type 2 Diabetes Mellitus patient education brochure in PDF format). Control group participants will also be able to enter and view their basic self-monitoring data (such as blood glucose values), but they will not receive the structured, nurse-led DSMES intervention, interactive counseling, or tailored motivational support.

Outcome assessments will be conducted at baseline and at the end of the 12-week intervention period. Primary outcomes will include changes in diabetes self-management behaviors and glycemic control, assessed using a validated Type 2 diabetes self-management scale and laboratory measures such as HbA1c and blood glucose values obtained from hospital records. Secondary outcomes will include changes in diabetes-related distress, measured with a validated diabetes distress scale, and user experience with the digital program, assessed with a mobile or digital application usability scale. Sociodemographic and clinical data will also be collected using standardized forms.

The study is planned as a single-blind design, in which participants are not informed of the specific group allocation (intervention versus active control), although they may recognize differences in the intensity of the digital support they receive. Data analysis will follow the principles of randomized controlled trials, and appropriate statistical methods will be used to compare changes in outcomes between groups, controlling for baseline values.

The findings of this study are expected to contribute to the evidence base on digital, nurse-led DSMES interventions for young adults with T2DM. If effective, the program may inform future integration of structured digital education and support into routine diabetes care and may help improve clinical and psychosocial outcomes in this vulnerable age group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years.
* Diagnosis of Type 2 Diabetes Mellitus.
* Able to read and write in the study language.
* Has access to the internet and to a digital device (such as a smartphone, tablet, or computer).
* No communication barriers (e.g., hearing, speech, or severe cognitive impairment that would prevent understanding of the intervention and questionnaires).
* No physical or mental health condition that, in the opinion of the investigators, would prevent participation in the digital intervention and follow-up.
* Willing and able to use a digital platform/application for diabetes self-management education and support.
* Provides informed consent to participate in the study.

Exclusion Criteria:

* Diagnosis of Type 1 Diabetes Mellitus or gestational diabetes.
* Advanced diabetic retinopathy or other severe visual impairment that significantly limits the ability to use digital devices or read educational materials.
* Severe psychiatric disorder or cognitive impairment that would interfere with participation in the intervention or completion of study assessments.
* Any condition that the investigators judge to make the person unsuitable for participation (e.g., severe acute illness, terminal condition).
* Unwillingness or inability to use the digital platform or to share necessary clinical data for the purposes of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-06-16 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Diabetes Self-Management Behaviors | Baseline and at 12 weeks after the start of the intervention
  Diabetes self-management behaviors will be assessed using a validated Type 2 Diabetes self-management scale and the ADCES7™ self-care behavior assessment forms. The primary outcome is the change in total self-management score from baseline to the end of the 12-week intervention, comparing the intervention and active control groups.
Change in HbA1c | Baseline and at 12 weeks after the start of the intervention
  Glycemic control will be evaluated using glycated hemoglobin (HbA1c) values obtained from hospital laboratory records. The primary outcome is the change in HbA1c (%) from baseline to 12 weeks, comparing the intervention and active control groups.
Change in Diabetes Distress | Baseline and at 12 weeks after the start of the intervention
  Diabetes-related distress will be assessed using a validated Diabetes Distress Scale (DDS). The primary outcome is the change in total diabetes distress score from baseline to 12 weeks, comparing the intervention group receiving the digital nurse-led DSMES program with the active control group receiving usual care plus standard digital education.

CONTACTS AND LOCATIONS:
Overall Officials: HİCRAN BEKTAŞ, PROF. DR., Study Chair — Akdeniz University Faculty of Nursing
Locations (1):
- Van Regional Training and Research Hospital, Endocrinology and Metabolism Clinic, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study is a single-center doctoral thesis conducted within a hospital setting and is subject to institutional and ethics committee restrictions on sharing identifiable or potentially re-identifiable clinical data. Aggregated results will be reported in publications and presentations, but raw individual-level data will not be made publicly available.

DOCUMENTS (1):
  • Study Protocol (2026-01-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT07325838/Prot_000.pdf